CLINICAL TRIAL: NCT02436057
Title: Development and Validation of the Automated Evaluation of Gastrointestinal Symptoms (AEGIS) Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of California, Los Angeles (Other); VA Medical Center-West Los Angeles (U.S. Federal Agency); University of Michigan (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Brennan Spiegel, Professor-in-Residence of Medicine and Public Health, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0023; 7U01AR057936-05 (NIH)
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Abdominal Pain; Deglutition Disorders; Fecal Incontinence; Nausea; Diarrhea; Constipation; Gastroesophageal Reflux
MeSH Terms: conditions — Abdominal Pain; Deglutition Disorders; Fecal Incontinence; Nausea; Diarrhea; Constipation; Gastroesophageal Reflux

ARMS (2):
- Usual care (No Intervention): Individuals in this arm will undergo usual care with their physician.
- AEGIS (Automated Evaluation of Gastrointestinal Symptoms) (Experimental): Individuals in the AEGIS arm will be invited to use AEGIS/My GI Health prior to their clinic visit. For those who complete AEGIS/My GI Health, their physician will have access to their AEGIS symptom report (includes a GI symptom heat map and GI history) and tailored education prescription.
  Interventions: Other: AEGIS (Automated Evaluation of Gastrointestinal Symptoms)

INTERVENTIONS:
Other: AEGIS (Automated Evaluation of Gastrointestinal Symptoms)
  Arms: AEGIS (Automated Evaluation of Gastrointestinal Symptoms)

SUMMARY:
Through a four-year grant awarded to the University of California at Los Angeles in 2009, Dr. Brennan Spiegel served as a principal investigator (PI) for a project to develop and initially validate a bank of items to assess gastrointestinal (GI) symptoms for the National Institutes of Health's (NIH's) Patient Reported Outcomes Measurement Information System (PROMIS). By the end of the grant period in July 2013, the project team had successfully developed and initially validated eight scales measuring the most common GI symptoms.

Afterwards, Dr. Spiegel's PROMIS team joined forces with the UCLA Computing Technology Research Laboratory (CTRL) and the University of Michigan Center for Healthcare Communication Research to develop the Automated Evaluation of Gastrointestinal Symptoms (AEGIS) algorithm which is delivered via My GI Health, an open--source Internet based patient-provider portal (P3) designed to enhance the delivery of GI health care (www.MyGIHealth.org). Through My GI Health and AEGIS, patients are able to complete PROMIS GI symptom measures and provide additional information about their GI symptoms and histories from computers, tablets or smart phones without the constraints of physical locale. This information is condensed into a GI PROMIS scores report and initial GI history that patients' providers can review prior to or concurrent with seeing the patient. The report, which can be incorporated into the electronic health record (EHR), helps busy clinicians to quickly understand the patient's complaints, document their symptoms and GI history, and leaves more time for conversation with the patient.

Beyond focusing their interaction, My GI Health also supports both the clinician and patient with an individualized "educational prescription" which guides the patient through a library of multi-media educational materials on GI symptoms, conditions, and treatments also contained within the website. The prescription is initially created by the website based on each patient's unique GI PROMIS "fingerprint", and can be modified by the provider based on their interaction with the patient. The clinician and patient can also access the PROMIS-tailored education in the exam room to jointly review pertinent materials, including animations of normal and abnormal GI functions, further reinforcing the patients' educational experiences around the PROMIS symptoms.

The aim of this current study is to validate the use of GI PROMIS in clinical practice by conducting a pragmatic clinical trial (PCT) comparing delivery of GI PROMIS on a novel e--platform vs. usual care.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the gastrointestinal clinic for evaluation.
* Able to read and write English.
* Has basic computing skills.

Exclusion Criteria:

* Having been seen and evaluated in the gastrointestinal clinic within the last 8 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | CG-CAHPS completed within 2 months of their clinic visit
  The Consumer Assessment of Health Providers & Systems Clinician and Group Survey - Adult Visit Questionnaire 2.0 (CG-CAHPS) will be used to assess patient satisfaction.

SECONDARY OUTCOMES:
Patient Assessment of Physician Interpersonal Skills | DISQ completed within 2 months of their clinic visit
  The Doctors' Interpersonal Skills Questionnaire (DISQ) will be used to assess patient assessment of physician interpersonal skills.
Patient Assessment of Shared Decision Making | SDM-Q-9 completed within 2 months of their clinic visit
  The 9-item Shared Decision Making Questionnaire (SDM-Q-9) will be used to assess patient assessment of shared decision making.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - West Los Angeles VA Medical Center, Los Angeles, California
  - University of Michigan, Ann Arbor, Michigan